CLINICAL TRIAL: NCT07014033
Title: Single-use Versus Multiple-use Endoscopes in Gastroenterology: Multi Methods Analysis to Balancing Infection Control and Environmental Impact
Brief Title: Single-use Versus Multiple-use Endoscopes in Gastroenterology
Acronym: SUMU-Endo
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RA627423; 24/PR/0316 (Other: Research Ethics Commmittee)
Record Dates: First submitted 2025-05-12; First posted 2025-06-10 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Endoscopy, Gastrointestinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who have recieved an Upper GI endoscopy
- Staff: Staff working in the endoscopy pathway

SUMMARY:
Gastroenterology is a branch of medicine that looks after people with problems in the gut (including the stomach and bowels) using an endoscope. An endoscope is a thin tube with a light and camera at the end, which is used to look inside bits of the body, for example the stomach, bile ducts (tubes that connect the liver and gallbladder to the bowel) or large bowel. Some have extra bits attached to take samples of tissue to look at under a microscope. These tubes are made mostly of plastic.

Around 1.5 million endoscopies are performed each year in the UK. In the NHS, most endoscopes are re-usable and are used hundreds of times after cleaning and disinfection. They must be very carefully cleaned and disinfected to reduce the risk of passing on infections to other patients as well as the healthcare staff who use the equipment. If endoscopes are cleaned and disinfected properly, the risk of infection will be very low. However there have been reports of infections, which may be related to disinfection not being done properly. Disposable single-use endoscopes are now available, designed to reduce the risk of infection. These are thought to be just as good as re-usable endoscopes. However, if we switch to disposable endoscopes, it may increase the cost to the NHS. There will also be an effect on the environment from using limited resources to make endoscopes, and get rid of them by incineration (burning) or burial in landfill waste.

The aim of this research is to provide evidence on the arguments for and against the use of single-use vs. multiple-use endoscopes in gastroenterology for NHS decision makers, especially regarding cost-effectiveness and effect on the environment. This will help the aim of the NHS in England to be "the world's first 'net zero' national health service.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Over the age of 18
* Patient has been invited to an NHS endoscopic clinic to undertake an upper GI endoscope procedure, including diagnostic endoscopies and the less complex therapeutic endoscopy.
* Patient is able to read and understand information provided
* Patient has capacity to provide consent
* Patient is able to participate in an interview. Staff
* Over the age of 18
* Employed by the NHS
* Working in relevant endoscopy unit - primary work involves the conduct of endoscopy and/or waste disposal services (decontamination or disposal).

Exclusion Criteria:

* Patient has received a lower GI endoscopy, e.g. colonoscopy or sigmoidoscopy
* Non-NHS service providers and receivers. (e.g., private diagnostic clinics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have attended or are scheduled to attend the endoscopy clinic at selected hospital sites.
  Staff who work in the endoscopy pathway: doctors/nurses, decontamination technicians etc.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative interview study | From recruitment to end of interview.
  As this is a qualitative interview study, there is no formal outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Coventry and Warwickshire NHS Trust, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided